CLINICAL TRIAL: NCT02512991
Title: Helicopter Versus Ground Emergency Medical Systems and the Effect on Mortality and Labour Market Affiliation of Patients Bound for Percutaneous Coronary Intervention
Brief Title: Follow-up of Patients Bound for PCI After Implementation of a Helicopter Emergency Medical System
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Kamilia S. Funder, MD., Rigshospitalet, Denmark
Other Study IDs: ALH2-KF-2015
Record Dates: First submitted 2015-07-27; First posted 2015-07-31 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: ST-elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HEMS patients: Patients bound for Percutaneous Coronary Intervention (PCI) at the PCI centre at Copenhagen University Hospital, Rigshospitalet, and who were transported by Helicopter Emergency Medical Service (HEMS) in a 36-month period (May 1st 2010 - April 30th 2013).
  Interventions: Other: Helicopter Emergency Medical Service
- GEMS patients: Patients bound for Percutaneous Coronary Intervention (PCI) at the PCI centre at Copenhagen University Hospital, Rigshospitalet, and who were transported by Ground Emergency Medical Service in a 40-month period (January 1st 2010 - April 30th 2013).

INTERVENTIONS:
Other: Helicopter Emergency Medical Service — May 1st 2010, the first Danish Helicopter Emergency Medical System (HEMS) was implemented in Region Zealand and the Capital Region of Denmark.
  Groups: HEMS patients

SUMMARY:
This study compares patients bound for Percutaneous Coronary Intervention (PCI) who were transported by either ground ambulance or emergency medical helicopter. The investigators describe long-term follow-up in relation to mortality and labour affiliation.

DETAILED DESCRIPTION:
Since 2003, percutaneous coronary intervention (PCI) for ST-Segment elevation myocardial infarction (STEMI) has been the preferred therapy in Denmark over fibrinolysis (thrombolysis) if performed within 120 minutes. Nevertheless, centralisation of designated PCI-centres may lead to systems delays as transport distance may be longer instead of just choosing thrombolysis at the nearest hospital.

As every minute counts when trying to minimize the ischemic injury and size of infarction following an acute coronary event, timely transportation by helicopter may facilitate overall prognosis.

As a part of a national initiative to improve prehospital care of patients with time critical illness such as myocardial infarction (MI), the first Danish Helicopter Emergency Medical System (HEMS) was implemented in the eastern part of Denmark May 1st 2010.

An initial study on 450 patients investigating short-term effects, found that HEMS significantly reduced time from the first electrocardiogram (ECG) diagnosis on-scene to arrival at the cardiac catheterisation laboratory (CCL) despite longer transport distances. Investigators also found a lower, but insignificant 30-day mortality in HEMS patients, adjusted OR=0.40 (95% CI=0.12-1.39, p=0.14).

The aim of the present study is to investigate long-term effects of HEMS in relation to mortality and labour market affiliation.

ELIGIBILITY:
Inclusion Criteria:

* The investigators include all STEMI patients having acute coronary angiography performed at the PCI centre at Copenhagen University Hospital, Rigshospitalet in a 40-month period from January 1st 2010 until April 30th 2013; and who were diagnosed with STEMI within the geographical area covered by both HEMS and GEMS. Patients with multiple contacts; only first contact is eligible.

Exclusion Criteria:

* The investigators exclude patients with cardiac arrest before hospital admission. For labour market analyses the investigators exclude patients not working full time three weeks prior to admission.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All STEMI patients having acute coronary angiography performed at the PCI centre at Copenhagen University Hospital, Rigshospitalet in a 40-month period from January 1st 2010 until April 30th 2013; and who were diagnosed with STEMI within the geographical area covered by both HEMS and GEMS.
  Patients are divided into two groups: 1) "field triaged" (ECG recorded out-of-hospital) and 2) inter-hospital transfers (ECG recorded in-hospital).
Sampling Method: Probability Sample
Enrollment: 1604 (Actual)
Dates: Start 2010-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Short term mortality after admission to the PCI unit | 30 day mortality

SECONDARY OUTCOMES:
Long-term mortality after admission to the PCI unit. | Mortality up to 5.5 years after admission to the PCI-unit
1-year mortality after admission to the PCI unit. | 1-year mortality
Time to involuntary early retirement or death from any cause | Up to 5.5 years after admission to the PCI unit
Reduced work ability two years after the coronary event (yes/no). | Two years after admission to the PCI unit
Time on social transfer payments during the first two years after the coronary event | Two years after admission to the PCI unit
Time to involuntary early retirement | Up to 5.5 years after admission to the PCI unit

CONTACTS AND LOCATIONS:
Overall Officials: Kamilia Funder, MD, Principal Investigator — Department of Anaesthesia, HOC 4231, Rigshospitalet

REFERENCES:
- [Background] Hesselfeldt R, Pedersen F, Steinmetz J, Vestergaard L, Simonsen L, Jorgensen E, Clemmensen P, Rasmussen LS. Implementation of a physician-staffed helicopter: impact on time to primary PCI. EuroIntervention. 2013 Aug 22;9(4):477-83. doi: 10.4244/EIJV9I4A77. PMID 23965353
- [Background] Laut KG, Hjort J, Engstrom T, Jensen LO, Tilsted Hansen HH, Jensen JS, Pedersen F, Jorgensen E, Holmvang L, Pedersen AB, Christensen EF, Lippert F, Lang-Jensen T, Jans H, Hansen PA, Trautner S, Kristensen SD, Lassen JF, Lash TL, Clemmensen P, Terkelsen CJ. Impact of health care system delay in patients with ST-elevation myocardial infarction on return to labor market and work retirement. Am J Cardiol. 2014 Dec 15;114(12):1810-6. doi: 10.1016/j.amjcard.2014.09.018. Epub 2014 Sep 28. PMID 25438906
- [Background] Andersen HR, Nielsen TT, Rasmussen K, Thuesen L, Kelbaek H, Thayssen P, Abildgaard U, Pedersen F, Madsen JK, Grande P, Villadsen AB, Krusell LR, Haghfelt T, Lomholt P, Husted SE, Vigholt E, Kjaergard HK, Mortensen LS; DANAMI-2 Investigators. A comparison of coronary angioplasty with fibrinolytic therapy in acute myocardial infarction. N Engl J Med. 2003 Aug 21;349(8):733-42. doi: 10.1056/NEJMoa025142. PMID 12930925